CLINICAL TRIAL: NCT02013921
Title: Evaluation du Niveau d'activité Physique Quotidien, Chez Des Patientes Porteuses d'un Cancer du Sein en période Post thérapeutique
Brief Title: Interest of Daily Physical Activity After Cancer Treatment
Acronym: APQ
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I12040
Record Dates: First submitted 2013-11-25; First posted 2013-12-17 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2015-04

CONDITIONS: Cancer; Tiredness
Keywords: Physical activity; Cancer
MeSH Terms: conditions — Neoplasms; Fatigue; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Physical Activity: Patients with a breast cancer and are completing treatment
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity

SUMMARY:
Many studies have demonstrated the beneficial effects of Adapted Physical Activity (APA) in different cancer types.

It therefore seems necessary to assess spontaneous Physical Activity in order to integrate it to the overall calculation of physical activity in clinical practice.

To assess the AP, two types of methods are validated : the subjective method using a questionnaries and objective method using a pedometer , accelerometer or measures calorimetry .

Subjective method shows , good acceptability by patients and low cost but can sometimes lead to poor estimation of the level of activity.

Objective methods obviously increase the accuracy of assessments but are more difficult to use for epidemiological studies , less accepted by the patient and more expensive.

In this study the investigators will measure the spontaneous Daily Physical Activity by both methods andd evaluate the correclation.

ELIGIBILITY:
Inclusion Criteria:

* adult (age ≥ 18 years)
* Having been informed of the study orally and in writing and have not expressed opposition to his participation
* Performance status <2
* Invasive breast adenocarcinoma, histologically documented.
* Patients with a breast cancer and are completing treatment
* Exclusion Criteria:
* Patient with metastatic cancer.
* Patient for which monitoring required by the protocol is impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a breast cancer and are completing treatment
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Daily physical activity assessment at 3 months | Month 3
  Physical activity is measured by means of an Actigraph. Patients will measure their daily physical activity , three times during one week espaced by 1 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncologie- CHU Limoges, Limoges, France